CLINICAL TRIAL: NCT06857643
Title: Functional Outcome After Surgery for Cervical Disc Prolapse
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrahman Zakaria Abdelrahman, residant doctor, Assiut University
Other Study IDs: Functional Outcome CDH Surgery
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cervical Disc Herniation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cervical disc herniation: Patients with degenerative cervical disc prolapse. patients who are subjected to Anterior cervical discectomy and fusion for patients with CDH occupying less than 50% of cervical canal and combined posterior laminectomy and Anterior cervical discectomy and fusion for patients with CDH occupying 50% or more of the cervical canal with canal stenosis

SUMMARY:
Cervical disc herniation (CDH) is the result of the displacement of the nucleus pulposus of the intervertebral disc, which may result in impingement of the traversing nerves as they exit the neural foramen or directly compressing the spinal cord contained within the spinal canal.[1] Eventually symptoms may arise because of a CDH with compression of the rootlet or spinal cord.[2] When conservative treatment for CDH fails, surgical treatment may be considered.[3] The main goals of surgical treatment are to remove pressure from the nerves, restore the alignment of the vertebrae, to stabilize the spine [3] and to prevent progression of neurological deficit in case of myelopathy.[4] Anterior cervical discectomy and fusion (ACDF) has proven to be an effective surgical intervention for both cervical radiculopathy and myelopathy and has become standard treatment for both of these disease states over the last half century.[5] Certain reports have indicated that various complications are associated with ACDF namely, incomplete decompression, recurrence of myelopathy due to adjacent segment degeneration.[6] In cases where the stenosis is extensive, or attributed in part to congenital stenosis, the posterior approach may be advantageous to achieve more extensive decompression that would otherwise not be possible through an anterior approach.[7] Given that most stenosis occurs from anterior pathology, a posterior decompression works to indirectly relieve pressure on the spinal cord.[8] Misalignment and large anterior compression of the spinal cord can be risk factors for insufficient functional recovery in patients treated with posterior decompression alone.[9] In this study we will perform ACDF for patients with CDH occupying less than 50% of cervical canal and combined posterior laminectomy and ACDF for patients with CDH occupying 50% or more of the cervical canal with canal stenosis.Cervical disc herniation (CDH) is the result of the displacement of the nucleus pulposus of the intervertebral disc, which may result in impingement of the traversing nerves as they exit the neural foramen or directly compressing the spinal cord contained within the spinal canal.[1] Eventually symptoms may arise because of a CDH with compression of the rootlet or spinal cord.[2] When conservative treatment for CDH fails, surgical treatment may be considered.[3] The main goals of surgical treatment are to remove pressure from the nerves, restore the alignment of the vertebrae, to stabilize the spine [3] and to prevent progression of neurological deficit in case of myelopathy.[4] Anterior cervical discectomy and fusion (ACDF) has proven to be an effective surgical intervention for both cervical radiculopathy and myelopathy and has become standard treatment for both of these disease states over the last half century.[5] Certain reports have indicated that various complications are associated with ACDF namely, incomplete decompression, recurrence of myelopathy due to adjacent segment degeneration.[6] In cases where the stenosis is extensive, or attributed in part to congenital stenosis, the posterior approach may be advantageous to achieve more extensive decompression that would otherwise not be possible through an anterior approach.[7] Given that most stenosis occurs from anterior pathology, a posterior decompression works to indirectly relieve pressure on the spinal cord.[8] Misalignment and large anterior compression of the spinal cord can be risk factors for insufficient functional recovery in patients treated with posterior decompression alone.[9] In this study we will perform ACDF for patients with CDH occupying less than 50% of cervical canal and combined posterior laminectomy and ACDF for patients with CDH occupying 50% or more of the cervical canal with canal stenosis.

the aim of the study to Assessment of the functional outcome after surgery for cervical disc prolapse

DETAILED DESCRIPTION:
Cervical disc herniation (CDH) is the result of the displacement of the nucleus pulposus of the intervertebral disc, which may result in impingement of the traversing nerves as they exit the neural foramen or directly compressing the spinal cord contained within the spinal canal.[1] Eventually symptoms may arise because of a CDH with compression of the rootlet or spinal cord.[2] When conservative treatment for CDH fails, surgical treatment may be considered.[3] The main goals of surgical treatment are to remove pressure from the nerves, restore the alignment of the vertebrae, to stabilize the spine [3] and to prevent progression of neurological deficit in case of myelopathy.[4] Anterior cervical discectomy and fusion (ACDF) has proven to be an effective surgical intervention for both cervical radiculopathy and myelopathy and has become standard treatment for both of these disease states over the last half century.[5] Certain reports have indicated that various complications are associated with ACDF namely, incomplete decompression, recurrence of myelopathy due to adjacent segment degeneration.[6] In cases where the stenosis is extensive, or attributed in part to congenital stenosis, the posterior approach may be advantageous to achieve more extensive decompression that would otherwise not be possible through an anterior approach.[7] Given that most stenosis occurs from anterior pathology, a posterior decompression works to indirectly relieve pressure on the spinal cord.[8] Misalignment and large anterior compression of the spinal cord can be risk factors for insufficient functional recovery in patients treated with posterior decompression alone.[9] In this study we will perform ACDF for patients with CDH occupying less than 50% of cervical canal and combined posterior laminectomy and ACDF for patients with CDH occupying 50% or more of the cervical canal with canal stenosis.

the aim of the study to Assessment of the functional outcome after surgery for cervical disc prolapse

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative cervical disc prolapse.

Exclusion Criteria:

* Traumatic Cervical disc prolapse
* Patients with ossification of the posterior longitudinal ligament (OPLL)

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: atients with degenerative cervical disc prolapse who underwint ACDF for patients with CDH occupying less than 50% of cervical canal and combined posterior laminectomy and ACDF for patients with CDH occupying 50% or more of the cervical canal with canal stenosi
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement in The modified Japanese orthopedic association (mJOA) score | 3 months
  The modified Japanese Orthopaedic Association (mJOA) score is an investigator-administered tool used to evaluate neurological function in patients with DCM . It is an 18-point scale that addresses upper (5 points) and lower extremity (7 points) motor function, sensation (3 points) and micturition (3 points). A score of 18 reflects no neurological deficits whereas a lower score indicates a greater degree of disability and functional impairment. The mJOA is the second most commonly used outcome measure to quantify severity in patients with DCM